CLINICAL TRIAL: NCT01890746
Title: A Randomized, Blinded, Placebo-Controlled, Dose Finding Study to Assess the Safety and Efficacy of the Oral Thrombopoietin Receptor Agonist, Eltrombopag, Administered to Subjects With Acute Myelogenous Leukaemia (AML) Receiving Induction Chemotherapy
Brief Title: A Safety and Efficacy Study of Eltrombopag in Subjects With AML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 117146; 2013-000642-20 (EudraCT Number)
Record Dates: First submitted 2013-06-27; First posted 2013-07-02 (Estimated); Results first posted 2016-06-14 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-08

CONDITIONS: Acute Leukaemia
Keywords: AML; de novo AML; leukemia; sAML/MDS; acute myeloid leukemia; acute myelogenous leukemia (AML); secondary acute myeloid leukemia; ETB115; Eltrombopag; thrombocytopenia; oral thrombopoietin receptor agonist
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Thrombocytopenia | interventions — Daunorubicin; Cytarabine; eltrombopag

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Eltrombopag arm (Experimental): Subjects received induction chemotherapy consisting of daunorubicin bolus intravenous (IV) infusion on Days 1-3 + cytarabine continuous IV infusion on Days 1-7 followed by Eltrombopag once daily orally starting on Day 4 of initial induction chemotherapy. If platelet count was not greater than 100 Gi/L after 7 days the dose was increased until a platelet count of at least 200 Gi/L was achieved/until remission was assessed/ maximum of 42 days from the start of the chemotherapy induction. Subjects who were not aplastic after first cycle of induction chemotherapy received second induction chemotherapy with a modified daunorubicin dose on Days 1-3 + cytarabine on Days 1-7.
  Interventions: Drug: Daunorubicin; Drug: Cytarabine; Drug: Eltrombopag
- Placebo arm (Placebo Comparator): Subject received induction chemotherapy consisting of daunorubicin bolus IV infusion on Days 1-3 + cytarabine continuous IV infusion on Days 1-7 followed by matching placebo once daily oral dose starting on Day 4 of initial induction chemotherapy. If platelet count was not greater than 100 Gi/L after 7 days the matching placebo was given until a platelet count of at least 200 Gi/L was achieved/ until remission was assessed/ maximum of 42 days from the start of the chemotherapy induction. Subjects who were not aplastic after first cycle of induction chemotherapy received a second induction chemotherapy with a modified daunorubicin dose on Days 1-3 + cytarabine on Days 1-7.
  Interventions: Drug: Daunorubicin; Drug: Cytarabine; Drug: Placebo

INTERVENTIONS:
Drug: Daunorubicin — For subjects between the ages of 18 and 60 years, 90 mg/m2/day by bolus IV injection through a freshly established free-flowing IV line for 10-15 minutes on days 1, 2, and 3. For subjects > 60 years: daunorubicin dose was adjusted to 60mg /m2.
Drug: Cytarabine — 100 mg/m2/day continuous IV infusion on Days 1 through 7.
Drug: Eltrombopag — 200 mg orally, once daily, beginning on Day 4 of the first cycle of induction. After 7 days, the dose of the Investigational Product (IP) was to be increased to 300 mg if platelet counts were <100 Gi/L. IP continued until achievement of platelet count of at least 200 Gi/L or assessment of remission of bone marrow status or a maximum of 42 days after initiation of most recent induction. In subjects of East Asian heritage 100 mg orally once daily (a 50% dose reduction) was used and after 7 days, the dose of IP was increased to 150 mg if platelet counts were <100 Gi/L.
  Arms: Eltrombopag arm
Drug: Placebo — Orally, once daily, beginning on Day 4 of the first cycle of induction. After 7 days, the dose given was matching 300 mg Eltrombopag if platelet counts were <100 Gi/L. Placebo continued until achievement of platelet count of at least 200 Gi/L or assessment of remission of bone marrow status or a maximum of 42 days after initiation of most recent induction. In subjects of East Asian heritage placebo matching 100 mg Eltrombopag orally once daily was used and after 7 days, the placebo matching 150 mg Eltrombopag was given if platelet counts were <100 Gi/L.
  Arms: Placebo arm

SUMMARY:
The purpose of this randomized, blinded, placebo-controlled study was to provide clinical safety and exploratory efficacy data on the use of Eltrombopag in adult subjects with Acute Myeloid Leukemia (AML) receiving standard induction chemotherapy with daunorubicin plus cytarabine. A minimum of 120 evaluable subjects newly diagnosed with AML was stratified by antecedent malignant hematologic disorder and age.

ELIGIBILITY:
Inclusion Criteria

* Age >=18 years
* Diagnosed with AML according to the WHO 2008 classification. Note: subjects with secondary AML following Myelodysplastic syndrome or secondary to previous leukemogenic therapy are allowed provided that a record of previous MDS history or leukemogenic therapy history is available.
* Eligible for induction by daunorubicin + cytarabine.
* Eligible to give informed consent to participate in the study.
* Have adequate baseline organ function defined by the following criteria:

Total bilirubin <=1.5 x upper limit of normal (ULN) except for Gilbert's syndrome, or other conditions that are not indicative of inadequate liver function (i.e. elevation of indirect bilirubin (haemolytic) in the absence of alanine aminotransferase [ALT] abnormality).

ALT <=3 x ULN. Serum Creatinine <=2.5 x ULN.

* Adequate cardiac function with LVEF >=50% as assessed by echocardiogram (ECHO) or Multi Gated Acquisition Scan (MUGA.
* Subjects with a QT interval corrected for heart rate according to Bazett's formula (QTcB) <450millisecond (msec) or <480msec for subjects with bundle branch block. The QTc should be based on single or averaged QTc values of triplicate electrocardiograms (ECGs) obtained over a brief recording period.
* Women must be either of non-childbearing potential or women with child-bearing potential and men with reproductive potential must be willing to practice acceptable methods of birth control during the study.
* Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception from time of randomization until 30 days after the last dose of investigational product.
* Women of childbearing potential must have a negative serum pregnancy test within 7 days of first dose of study treatment and agree to use effective contraception during the study and for 30 days following the last dose of investigational product.

Exclusion Criteria

* A diagnosis of acute promyelocytic (M3) or acute megakaryocytic leukaemia (M7).
* Previous history of exposure to an anthracycline compound.
* Previous AML treatment (other than hydroxyurea).
* Any serious medical condition, laboratory abnormality, or psychiatric illness that, in the view of the treating physician, would place the participant at an unacceptable risk if he or she were to participate in the study or would prevent that person from giving informed consent.
* History of thromboembolic event or other condition requiring ongoing use of anticoagulation either with warfarin or low molecular-weight heparin. Note: Occlusion of a central line is not exclusion.
* Treatment with an investigational drug within 30 days or 5 half lives, whichever is longer, preceding the first dose of study medication.
* Current and continued use during study treatment period of known Breast cancer resistance protein (BCRP) inhibitors or known P-gp inhibitors.
* Known active hepatitis B, hepatitis C or Human Immunodeficiency Virus (HIV) infection.
* Known hypersensitivity to any of the study drugs or its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2013-09-05 (Actual); Primary Completion 2015-03-13 (Actual); Study Completion 2017-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (40):
- United States (14):
  - Novartis Investigative Site, Farmington, Connecticut
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Ames, Iowa
  - Novartis Investigative Site, Sioux City, Iowa
  - Novartis Investigative Site, Burlington, Massachusetts
  - Novartis Investigative Site, Kansas City, Missouri
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Canton, Ohio
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Providence, Rhode Island
  - Novartis Investigative Site, Nashville, Tennessee
- Australia (3):
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Parkville, Victoria
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
- Canada (2):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Pátrai
- Hungary (2):
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Szeged
- Israel (5):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Holon
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Tel Aviv
- Poland (2):
  - Novartis Investigative Site, Słupsk
  - Novartis Investigative Site, Wroclaw
- Russia (6):
  - Novartis Investigative Site, Kaluga
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Penza
  - Novartis Investigative Site, St'Petersburg
  - Novartis Investigative Site, Tula
- South Korea (2):
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Seoul, Korea

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Frey N, Jang JH, Szer J, Illes A, Kim HJ, Ram R, Chong BH, Rowe JM, Borisenkova E, Liesveld J, Winer ES, Cherfi A, Aslanis V, Ghaznawi F, Strickland S. Eltrombopag treatment during induction chemotherapy for acute myeloid leukaemia: a randomised, double-blind, phase 2 study. Lancet Haematol. 2019 Mar;6(3):e122-e131. doi: 10.1016/S2352-3026(18)30231-X. Epub 2019 Jan 29. PMID 30704923

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (Par.) diagnosed with Acute Myelogenous Leukemia (AML) of any subtype (except acute promyelocytic [M3] or acute megakaryocytic leukaemia [M7]) were eligible for the study.
Pre-assignment Details: Sufficient number of participants were screened and 148 participants were randomized and entered in to the study. Participants were stratified by antecedent malignant hematologic disorder (yes versus no) and age (18-60 years versus >60 years), before they were randomized to receive study treatments.
Groups:
- Eltrombopag (ELQ) QD: Par. received IDN CTY consisting of DAU bolus IV INF on D 1-3 at a dose of 90 mg/m^2 for Par. 18-60 years old or 60 mg/m^2 for Par.>60 years old plus cytarabine 100 mg/m^2 continuous IV INF on D1-7. Par. received ELT as 200 mg (100 mg for East-Asian Heritage) QD oral dose starting on D4 of initial IDN CTY at least 20 hours after end of D3 DAU INF. If PT count was not >100 Gi/L after 7 days the dose was increased to 300 mg (150 mg East-Asian Heritage) QD until a PT count of at least 200 Gi/L was achieved, until remission was assessed by bone marrow biopsy, or for a maximum of 42 days from the start of the CTY IDN cycle. Par. who were not aplastic after first cycle of IDN CTY received re-IDN with a modified DAU dose of 45mg/m^2/day on D1-3 plus cytarabine 100 mg/m^2/day on D1-7. For re-IDN Par., ELT was held from D1-3 of re-IDN, and resumed on D4 at the same dose and duration.
- Placebo QD: Participants received first line IDN CTY consisting of DAU bolus IV INF on Days 1-3 at a dose of 90 mg/m^2 for participants 18-60 years old or 60 mg/m^2 for participants >60 years of age plus cytarabine continuous IV INF on Days 1-7 at a dose of 100 mg/m^2. Participants received placebo QD oral dose starting on Day 4 of initial IDN CTY at least 20 hours after end of Day 3 DAU INF up to a maximum duration of 42 days.
Period: Overall Study
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Started | 74 | 74
Completed | 22 | 33
Not Completed | 52 | 41
Not completed — Death | 39 | 30
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 4 | 1
Not completed — Physician Decision | 3 | 2
Not completed — Withdrawal by Subject | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD | Total
Number analyzed (Participants) | 74 | 74 | 148
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The Intent-to-Treat (ITT) population comprised all randomized subjects regardless of whether or not study treatment was administered.
  Years | 56.7 (12.25) | 56.6 (11.58) | 56.7 (11.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 31 | 69
  Male | 36 | 43 | 79
Race/Ethnicity, Customized [Number; unit: Participants] — Population: The Intent-to-Treat (ITT) population comprised all randomized subjects regardless of whether or not study treatment was administered.
  Participants
    African American/African Heritage | 1 | 2 | 3
    Asian - Central/South Asian Heritage | 0 | 1 | 1
    Asian - East Asian Heritage | 26 | 17 | 43
    Asian - South East Asian Heritage | 0 | 1 | 1
    White - Arabic/North African Heritage | 5 | 3 | 8
    White - White/Caucasian/European Heritage | 42 | 50 | 92

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Events (AE) and Any Serious Adverse Events (SAE) as a Measure of Safety and Tolerability.
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, is an important medical event that jeopardizes the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition, or is associated with liver injury and impaired liver function.
Time Frame: From the time the first dose of study treatment was administered until 30 days following discontinuation of investigational product regardless of initiation of a new cancer therapy or transfer to hospice
Population: Safety population: all subjects who received at least one dose of investigational product.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 71
Participants
  Any AE | 72 | 66
  Any SAE | 24 | 14

2. Primary Outcome: Change From Baseline in the Left Ventricular Ejection Fraction (LVEF).
Description: LVEF is a measurement of the percentage of blood leaving heart each time it contracts. LVEF was assessed by an echocardiogram (ECHO) or Multiple Gated Acquisition scan (MUGA). Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date. Change from Baseline was calculated as the Day 42 value minus the Baseline value.
Time Frame: Baseline and Day 42 of the latest chemotherapy cycle (Up to 8 weeks)
Population: Participants in the Safety Population who provided Baseline and Day 42 LVEF measurements.
Measure: Mean (Standard Deviation); unit: LVEF percent
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 71
LVEF percent
  chnge from baseline (BL) to end of study: number analyzed (Participants) | 57 | 62
  chnge from baseline (BL) to end of study | -2.5 (7.81) | -4.3 (8.54)
  change from BL to worse post-BL case: number analyzed (Participants) | 58 | 63
  change from BL to worse post-BL case | -4.1 (8.61) | -5.7 (9.05)

3. Primary Outcome: Number of Participants With Worst-case Grade Changes From Baseline in the Hematology Parameters
Description: The number of participants with a maximum post-baseline grade increase of Grade 3 (G3) or Grade 4 (G4) from their baseline grade are presented. Hematology parameters included only lab tests that are gradable by Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
Time Frame: Baseline and up to Day 42 of the latest chemotherapy cycle (Up to 8 weeks)
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 71
Participants
  Hemoglobin Low, G3 | 53 | 46
  Leukocytes, G3 | 10 | 10
  Leukocytes, G4 | 9 | 5
  Lymphocytes Low, G3 | 31 | 26
  Lymphocytes Low, G4 | 35 | 38
  Neutrophils, G4 | 44 | 39
  Platelets, G3 | 1 | 0
  Platelets, G4 | 63 | 56

4. Primary Outcome: Number of Participants With Worst-case Grade Changes From Baseline in the Clinical Chemistry Parameters
Description: The number of participants with a maximum post-baseline grade increase of Grade 3 or Grade 4 from their baseline grade are presented. Clinical Clinical Chemistry parameters included only lab tests that are gradable by CTCAE v4.0.
Time Frame: Baseline and up to Day 42 of the latest chemotherapy cycle (Up to 8 weeks)
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 71
Participants
  Alanine Aminotransferase, G3 | 1 | 5
  Albumin, G3 | 6 | 4
  Aspartate Aminotransferase, G3 | 0 | 1
  Bilirubin, G3 | 1 | 4
  Bilirubin, G4 | 0 | 1
  Calcium Low, G3 | 0 | 1
  Creatinine, G3 | 0 | 1
  Creatinine, G4 | 1 | 0
  Glucose High, G3 | 6 | 3
  Glucose High, G4 | 0 | 1
  Magnesium Low, G3 | 0 | 1
  Magnesium High, G3 | 3 | 0
  Phosphate, G3 | 10 | 19
  Phosphate, G4 | 1 | 0
  Potassium Low, G3 | 8 | 10
  Potassium Low, G4 | 0 | 2
  Potassium High, G3 | 4 | 0
  Potassium High, G4 | 1 | 1
  Sodium Low, G3 | 3 | 4
  Urate, G4 | 3 | 0

5. Primary Outcome: Number of Participants With Liver Events.
Description: The number of participants with liver enzyme (ALT, AST, ALP, Total bilirubin) abnormalities while receiving study treatment in each arm are presented.
Time Frame: 8 weeks
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 71
Participants | 2 | 6

6. Primary Outcome: Number of Participants With Worst-case Changes From Baseline in Electrocardiogram (ECG) Values
Description: The number of participants with worst case post-baseline changes (normal, abnormal - not clinically significant [NCS], abnormal - clinically significant [NS]) in ECG QT prolonged values are presented. The protocol does not define the criteria for normal, abnormal-NCS and abnormal CS ECG. The outcome was based solely on the investigator interpretation of ECG tracings.
Time Frame: Baseline and Day 42 of the latest chemotherapy cycle (Up to 8 weeks)
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 71
Participants
  Normal: number analyzed (Participants) | 59 | 63
  Normal | 34 | 33
  Abnormal - NCS: number analyzed (Participants) | 59 | 63
  Abnormal - NCS | 23 | 29
  Abnormal - CS: number analyzed (Participants) | 59 | 63
  Abnormal - CS | 2 | 1

7. Primary Outcome: Number of Participants With Worst-case Changes From Baseline in the Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: The number of participants with worst case post-baseline changes (improved, no change, deteriorated) are presented.
Time Frame: Baseline and Day 42 of the latest chemotherapy cycle (Up to 8 weeks)
Population: Participants in the Safety Population who provided Baseline and post-Baseline assessments.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 71
Participants
  Deteriorated | 36 | 36
  Improved | 0 | 1
  No Change | 37 | 34

8. Primary Outcome: Worst-case Change From Baseline in Pulse Rate Values
Description: The worst-case post Baseline high and low changes in pulse rate values from Baseline are presented. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date. Post Baseline is defined as the highest and lowest non-missing post Baseline value respectively. Change from Baseline was calculated as the post Baseline value minus the Baseline value.
Time Frame: Baseline and up to Day 42 of the latest chemotherapy cycle (Up to 8 weeks)
Population: Safety population. Only those participants available at the indicated time points were analyzed (represented by n=X, X in the category titles)
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 71
Beats/minute
  High: number analyzed (Participants) | 66 | 67
  High | 18.48 (20.616) | 17.73 (15.112)
  Low: number analyzed (Participants) | 61 | 55
  Low | -10.36 (14.039) | -11.24 (12.123)

9. Primary Outcome: Worst-case Post Baseline Change in Blood Pressure Values From Baseline
Description: The worst-case post Baseline high changes in systolic blood pressure (SBP) and diastolic blood pressure (DBP) values from Baseline are presented. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date. Change from Baseline was calculated as the visit value minus the Baseline value.
Time Frame: Baseline and up to Day 42 of the latest chemotherapy cycle (Up to 8 weeks)
Population: Safety population
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 71
millimeter of mercury (mmHg)
  SBP | 14.59 (17.936) | 14.34 (14.626)
  DBP | 9.38 (12.000) | 12.61 (10.947)

10. Primary Outcome: Worst-case Post Baseline Change in Temperature Values From Baseline
Description: The worst-case post Baseline high and low changes in temperature values from Baseline are presented. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date. Post Baseline was defined as the highest and lowest non-missing post Baseline value respectively. Change from Baseline was calculated as the post Baseline value minus the Baseline value.
Time Frame: Baseline and up to Day 42 of the latest chemotherapy cycle (Up to 8 weeks)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 71
Degrees Celsius
  High: number analyzed (Participants) | 70 | 69
  High | 0.62 (0.941) | 0.77 (0.879)
  Low: number analyzed (Participants) | 47 | 43
  Low | -0.44 (0.628) | -0.63 (0.592)

11. Secondary Outcome: Plasma Pharmacokinetics (PK) Parameter of Daunorubicin: Half-life (t1/2)
Description: Daunorubicin half-life. PK analyses used actual relative time and actual dosing information in mg/m2. All parameter values were divided by daunorubicin dose in mg/m2 except t1/2.
Time Frame: Cycle 1 Day 3 to Day 9 (0 to 144 hrs post-dose)
Population: PK population: The PK population consisted of all subjects who completed initial induction treatment and had at least 1 non-baseline blood sample for PK obtained and analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: hour (h)
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 72
hour (h) | 15.754 [13.969 to 17.766] | 13.709 [12.103 to 15.527]
Statistical Analysis 1: Comparison: Eltrombopag (ELQ) QD vs Placebo QD; Test type: Other — Bioequivalence; Ratio of geometric means (%) = 114.9, 90% CI 2-sided [99.5 to 132.7]

12. Secondary Outcome: Plasma Pharmacokinetics (PK) Parameter of Daunorubicinol: Half-life (t1/2)
Description: Daunorubicinol half-life. PK analyses used actual relative time and actual dosing information in mg/m2. All parameter values were divided by daunorubicin dose in mg/m2 except t1/2.
Time Frame: Cycle 1 Day 3 to Day 9 (0 to 144 hrs post-dose)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: hour (h)
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 72
hour (h) | 22.735 [21.187 to 24.396] | 21.603 [20.232 to 23.067]
Statistical Analysis 1: Comparison: Eltrombopag (ELQ) QD vs Placebo QD; Test type: Other — Bioequivalence; Ratio of geometric means (%) = 105.2, 90% CI 2-sided [97.1 to 114.0]

13. Secondary Outcome: Daunorubicin Dose-normalized Plasma: AUC(0-∞)
Description: Daunorubicin AUC(0-∞). PK analyses used actual relative time and actual dosing information in mg/m2. All parameter values were divided by daunorubicin dose in mg/m2 except t1/2.
Time Frame: Cycle 1 Day 3 to Day 9 (0 to 144 hrs post-dose)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: (h*ug/ml)/(mg/m2)
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 72
(h*ug/ml)/(mg/m2) | 8.0807 [7.0672 to 9.2396] | 8.7880 [7.3893 to 10.451]
Statistical Analysis 1: Comparison: Eltrombopag (ELQ) QD vs Placebo QD; Test type: Other — Bioequivalence; Ratio of geometric means (%) = 92.0, 90% CI 2-sided [76.8 to 110.2]

14. Secondary Outcome: Daunorubicinol Dose-normalized Plasma: AUC(0-∞)
Description: Daunorubicinol AUC(0-∞). PK analyses used actual relative time and actual dosing information in mg/m2. All parameter values were divided by daunorubicin dose in mg/m2 except t1/2.
Time Frame: Cycle 1 Day 3 to Day 9 (0 to 144 hrs post-dose)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: (h*ug/ml)/(mg/m2)
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 72
(h*ug/ml)/(mg/m2) | 63.997 [58.686 to 69.746] | 62.835 [58.673 to 67.292]
Statistical Analysis 1: Comparison: Eltrombopag (ELQ) QD vs Placebo QD; Test type: Other — Bioequivalence; Ratio of geometric means (%) = 101.8, 90% CI 2-sided [92.9 to 111.7]

15. Secondary Outcome: Daunorubicin Dose-normalized Plasma: AUC(24-∞)
Description: Daunorubicin AUC(24-∞). PK analyses used actual relative time and actual dosing information in mg/m2. All parameter values were divided by daunorubicin dose in mg/m2 except t1/2.
Time Frame: Cycle 1 Day 4 to Day 9 (24 to 144 hrs post-dose)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: (h*ug/ml)/(mg/m2)
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 72
(h*ug/ml)/(mg/m2) | 0.87496 [0.76202 to 1.0046] | 0.72315 [0.62633 to 0.83493]
Statistical Analysis 1: Comparison: Eltrombopag (ELQ) QD vs Placebo QD; Test type: Other — Bioequivalence; Ratio of geometric means (%) = 121.0, 90% CI 2-sided [102.5 to 142.8]

16. Secondary Outcome: Daunorubicinol Dose-normalized Plasma: AUC(24-∞)
Description: Daunorubicinol AUC(24-∞). PK analyses used actual relative time and actual dosing information in mg/m2. All parameter values were divided by daunorubicin dose in mg/m2 except t1/2.
Time Frame: Cycle 1 Day 4 to Day 9 (24 to 144 hrs post-dose)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: (h*ug/ml)/(mg/m2)
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 72
(h*ug/ml)/(mg/m2) | 24.537 [22.052 to 27.301] | 23.039 [21.169 to 25.074]
Statistical Analysis 1: Comparison: Eltrombopag (ELQ) QD vs Placebo QD; Test type: Other — Bioequivalence; Ratio of geometric means (%) = 106.5, 90% CI 2-sided [95.0 to 119.4]

17. Secondary Outcome: Daunorubicin Dose-normalized Plasma: AUC(0-t)
Description: Daunorubicin AUC(0-t). PK analyses used actual relative time and actual dosing information in mg/m2. All parameter values were divided by daunorubicin dose in mg/m2 except t1/2.
Time Frame: Cycle 1 Day 3 to Day 9 (0 to 144 hrs post-dose)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: (h*ug/ml)/(mg/m2)
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 72
(h*ug/ml)/(mg/m2) | 7.9523 [6.9485 to 9.1012] | 8.6723 [7.2855 to 10.323]
Statistical Analysis 1: Comparison: Eltrombopag (ELQ) QD vs Placebo QD; Test type: Other — Bioequivalence; Ratio of geometric means (%) = 91.7, 90% CI 2-sided [76.5 to 110.0]

18. Secondary Outcome: Daunorubicinol Dose-normalized Plasma: AUC(0-t)
Description: daunorubicinol AUC(0-t). PK analyses used actual relative time and actual dosing information in mg/m2. All parameter values were divided by daunorubicin dose in mg/m2 except t1/2.
Time Frame: Cycle 1 Day 3 to Day 9 (0 to 144 hrs post-dose)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: (h*ug/ml)/(mg/m2)
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 72
(h*ug/ml)/(mg/m2) | 62.463 [57.268 to 68.129] | 61.608 [57.500 to 66.009]
Statistical Analysis 1: Comparison: Eltrombopag (ELQ) QD vs Placebo QD; Test type: Other — Bioequivalence; Ratio of geometric means (%) = 101.4, 90% CI 2-sided [92.4 to 111.2]

19. Secondary Outcome: Daunorubicin Dose-normalized Plasma: AUC(24-t)
Description: Daunorubicin AUC(24-t). PK analyses used actual relative time and actual dosing information in mg/m2. All parameter values were divided by daunorubicin dose in mg/m2 except t1/2.
Time Frame: Cycle 1 Day 4 to Day 9 (24 to 144 hrs post-dose)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: (h*ug/ml)/(mg/m2)
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 72
(h*ug/ml)/(mg/m2) | 0.76524 [0.65947 to 0.88797] | 0.59660 [0.48882 to 0.72813]
Statistical Analysis 1: Comparison: Eltrombopag (ELQ) QD vs Placebo QD; Test type: Other — Bioequivalence; Ratio of geometric means (%) = 120.0, 90% CI 2-sided [100.7 to 142.6]

20. Secondary Outcome: Daunorubicinol Dose-normalized Plasma: AUC(24-t)
Description: Daunorubicinol AUC(24-t). PK analyses used actual relative time and actual dosing information in mg/m2. All parameter values were divided by daunorubicin dose in mg/m2 except t1/2.
Time Frame: Cycle 1 Day 4 to Day 9 (24 to 144 hrs post-dose)
Population: as for outcome 11
Measure: Geometric Mean (90% Confidence Interval); unit: (h*ug/ml)/(mg/m2)
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 72
(h*ug/ml)/(mg/m2) | 22.963 [20.557 to 25.651] | 21.821 [20.020 to 23.783]
Statistical Analysis 1: Comparison: Eltrombopag (ELQ) QD vs Placebo QD; Test type: Other — Bioequivalence; Ratio of geometric means (%) = 105.2, 90% CI 2-sided [93.6 to 118.3]

21. Secondary Outcome: Daunorubicin Dose-normalized Plasma: Cmax
Description: Daunorubicin Cmax. PK analyses used actual relative time and actual dosing information in mg/m2. All parameter values were divided by daunorubicin dose in mg/m2 except t1/2.
Time Frame: Cycle 1 Day 3 to Day 9 (0 to 144 hrs post-dose)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: (ug/ml)/(mg/m2)
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 72
(ug/ml)/(mg/m2) | 5.1527 [3.9561 to 6.7114] | 6.4113 [4.6773 to 8.7882]
Statistical Analysis 1: Comparison: Eltrombopag (ELQ) QD vs Placebo QD; Test type: Other — Bioequivalence; Ratio of geometric means (%) = 80.4, 90% CI 2-sided [57.2 to 113.0]

22. Secondary Outcome: Daunorubicinol Dose-normalized Plasma: Cmax
Description: Daunorubicinol Cmax. PK analyses used actual relative time and actual dosing information in mg/m2. All parameter values were divided by daunorubicin dose in mg/m2 except t1/2.
Time Frame: Cycle 1 Day 3 to Day 9 (0 to 144 hrs post-dose)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: (ug/ml)/(mg/m2)
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 72
(ug/ml)/(mg/m2) | 3.5770 [3.0433 to 4.2044] | 3.3640 [2.8433 to 3.9799]
Statistical Analysis 1: Comparison: Eltrombopag (ELQ) QD vs Placebo QD; Test type: Other — Bioequivalence; Ratio of geometric means (%) = 106.3, 90% CI 2-sided [87.6 to 129.0]

23. Secondary Outcome: Cycle 2: Daunorubicin Dose-normalized Plasma: AUC(0-24)
Description: Cycle 2 Daunorubicin AUC(0-24). PK analyses used actual relative time and actual dosing information in mg/m2. All parameter values were divided by daunorubicin dose in mg/m2 except t1/2.
Time Frame: Cycle 2 Day 1 to Day 2 (0 to 24 post-dose)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: (h*ug/ml)/(mg/m2)
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 10 | 12
(h*ug/ml)/(mg/m2) | 10.315 [6.7932 to 15.662] | 8.1146 [6.0221 to 10.934]
Statistical Analysis 1: Comparison: Eltrombopag (ELQ) QD vs Placebo QD; Test type: Other — Bioequivalence; Ratio of geometric means (%) = 127.1, 90% CI 2-sided [84.2 to 191.9]

24. Secondary Outcome: Cycle 2: Daunorubicinol Dose-normalized Plasma: AUC(0-24)
Description: Cycle 2 Daunorubicinol AUC(0-24). PK analyses used actual relative time and actual dosing information in mg/m2. All parameter values were divided by daunorubicin dose in mg/m2 except t1/2.
Time Frame: Cycle 2 Day 1 to Day 2 (0 to 24 post-dose)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: (h*ug/ml)/(mg/m2)
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 10 | 12
(h*ug/ml)/(mg/m2) | 34.067 [26.479 to 43.829] | 30.820 [24.148 to 39.335]
Statistical Analysis 1: Comparison: Eltrombopag (ELQ) QD vs Placebo QD; Test type: Other — Bioequivalence; Ratio of geometric means (%) = 110.5, 90% CI 2-sided [83.9 to 145.7]

25. Secondary Outcome: Cycle 2: Daunorubicin Dose-normalized Plasma: Cmax
Description: Cycle 2 Daunorubicin Cmax. PK analyses used actual relative time and actual dosing information in mg/m2. All parameter values were divided by daunorubicin dose in mg/m2 except t1/2.
Time Frame: Cycle 2 Day 1 to Day 2 (0 to 24 post-dose)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: (ug/ml)/(mg/m2)
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 10 | 12
(ug/ml)/(mg/m2) | 11.141 [4.3653 to 28.432] | 3.8905 [1.2805 to 11.820]
Statistical Analysis 1: Comparison: Eltrombopag (ELQ) QD vs Placebo QD; Test type: Other — Bioequivalence; Ratio of geometric means (%) = 286.4, 90% CI 2-sided [90.1 to 910.7]

26. Secondary Outcome: Cycle 2: Daunorubicinol Dose-normalized Plasma: Cmax
Description: Cycle 2 Daunorubicinol Cmax. PK analyses used actual relative time and actual dosing information in mg/m2. All parameter values were divided by daunorubicin dose in mg/m2 except t1/2.
Time Frame: Cycle 2 Day 1 to Day 2 (0 to 24 post-dose)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: (ug/ml)/(mg/m2)
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 10 | 12
(ug/ml)/(mg/m2) | 4.0200 [2.5302 to 6.3870] | 1.9868 [1.4247 to 2.7708]
Statistical Analysis 1: Comparison: Eltrombopag (ELQ) QD vs Placebo QD; Test type: Other — Bioequivalence; Ratio of geometric means (%) = 202.3, 90% CI 2-sided [131.3 to 311.8]

27. Secondary Outcome: Number of Platelet Transfusions Per Week Within Cycles
Description: This was the average number of platelet transfusions per week within cycles.
Time Frame: Post-Base line up to Day 42 of the latest chemotherapy cycle (Up to 8 weeks)
Population: The Intent-to-Treat (ITT) population comprised all randomized subjects regardless of whether or not study treatment was administered. This population was based on the treatment to which the subject was randomized.
Measure: Median (Standard Deviation); unit: Platelet transfusions per week
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 74
Platelet transfusions per week | 1.5 (1.18) | 1.4 (1.22)

28. Secondary Outcome: Time to Platelet Count Recovery >=20 Gi/L
Description: Time to Platelet counts >= 20 Gi/L for 3 consecutive days, unaided by transfusions in patients with < 20 Gi/L after chemotherapy. For this endpoint, the event required platelet count to be >= 20 Gi/L for 3 consecutive days. Hematology was assessed daily during hospital stay but only weekly after hospital discharge and thus, platelet count was not always available for 3 consecutive days to confirm the achievement of platelet count recovery.
Time Frame: From last dose of chemotherapy to up to end of study year 2 assessment
Population: as for outcome 27
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 70 | 68
Months | NA [NA to NA] — N/A = Not enough participants achieved platelet recovery >= 20 Gi/L | NA [NA to NA] — N/A = Not enough participants achieved platelet recovery >= 20 Gi/L
Statistical Analysis 1: Comparison: Eltrombopag (ELQ) QD vs Placebo QD; Test type: Superiority; p = 0.7461, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.28 to 2.48]

29. Secondary Outcome: Time to Platelet Recovery >=100 Gi/L
Description: Time to platelet counts >= 100 Gi/L unaided by transfusions in participants with < 100 Gi/L after chemotherapy.
Time Frame: From last dose of chemotherapy to up to end of study year 2 assessment
Population: as for outcome 27
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 73
Months | 0.69 [0.69 to 0.76] | 0.69 [0.69 to 0.82]
Statistical Analysis 1: Comparison: Eltrombopag (ELQ) QD vs Placebo QD; Test type: Superiority; p = 0.6175, Log Rank; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.74 to 1.63]

30. Secondary Outcome: Number of Participants Who Achieved Platelet Count Recovery by Day 21
Description: Number of participants with platelet counts 20 Gi/L for 3 consecutive days, unaided by transfusions, in patients with < 20 Gi/L after chemotherapy.
Time Frame: By Day 21
Population: as for outcome 27
Measure: Number; unit: Count of participants
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 70 | 68
Count of participants | 4 | 7
Statistical Analysis 1: Comparison: Eltrombopag (ELQ) QD vs Placebo QD; Test type: Superiority; p = 0.3224, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.5281, 95% CI 2-sided [0.1084 to 2.2086]

31. Secondary Outcome: Summary of Platelet Counts Over Time
Description: Platelet counts over time
Time Frame: Baseline, daily then weekly within cycle up to 42 days after last chemotherapy dose, end of therapy /remission assessment visit
Population: as for outcome 27
Measure: Median (Full Range); unit: Gi/L
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 74
Gi/L
  Baseline | 51.5 [5 to 241] | 50.0 [9 to 232]
  C1D1: number analyzed (Participants) | 59 | 66
  C1D1 | 52.0 [5 to 241] | 48.5 [9 to 232]
  C1D2 | 43.5 [4 to 237] | 42.0 [5 to 368]
  C1D3: number analyzed (Participants) | 72 | 72
  C1D3 | 35.5 [4 to 226] | 37.0 [7 to 220]
  C1D4: number analyzed (Participants) | 74 | 69
  C1D4 | 36.5 [3 to 227] | 29.0 [5 to 146]
  C1D5: number analyzed (Participants) | 73 | 71
  C1D5 | 33.0 [3 to 201] | 29.0 [5 to 146]
  C1D6: number analyzed (Participants) | 73 | 69
  C1D6 | 32.0 [4 to 164] | 30.0 [6 to 125]
  C1D7: number analyzed (Participants) | 73 | 70
  C1D7 | 27.0 [3 to 123] | 27.0 [4 to 102]
  C1D8: number analyzed (Participants) | 73 | 69
  C1D8 | 24.0 [2 to 99] | 22.0 [4 to 80]
  C1D9: number analyzed (Participants) | 72 | 69
  C1D9 | 20.5 [1 to 109] | 19.0 [5 to 59]
  C1D14: number analyzed (Participants) | 68 | 68
  C1D14 | 16.5 [0 to 70] | 18.0 [1 to 81]
  C1D21: number analyzed (Participants) | 51 | 55
  C1D21 | 39.0 [5 to 325] | 25.0 [2 to 232]
  C1D28: number analyzed (Participants) | 36 | 29
  C1D28 | 484.5 [14 to 1590] | 121.0 [7 to 539]
  C1D35: number analyzed (Participants) | 14 | 14
  C1D35 | 547.0 [15 to 1493] | 181.0 [10 to 424]
  C1D42: number analyzed (Participants) | 0 | 1
  C1D42 |  | 304.0 [304 to 304]
  C2D1: number analyzed (Participants) | 10 | 12
  C2D1 | 31.0 [12 to 1059] | 30.5 [10 to 432]
  C2D2: number analyzed (Participants) | 9 | 12
  C2D2 | 26.0 [3 to 831] | 28.5 [8 to 400]
  C2D3: number analyzed (Participants) | 10 | 12
  C2D3 | 25.5 [0 to 730] | 29.0 [8 to 437]
  C2D4: number analyzed (Participants) | 9 | 12
  C2D4 | 32.0 [2 to 678] | 35.5 [11 to 454]
  C2D5: number analyzed (Participants) | 10 | 11
  C2D5 | 37.0 [9 to 516] | 22.0 [12 to 476]
  C2D6: number analyzed (Participants) | 10 | 12
  C2D6 | 27.0 [4 to 430] | 33.0 [7 to 533]
  C2D7: number analyzed (Participants) | 7 | 12
  C2D7 | 24.0 [6 to 295] | 28.5 [12 to 390]
  C2D14: number analyzed (Participants) | 8 | 11
  C2D14 | 10.5 [3 to 31] | 16.0 [6 to 66]
  C2D21: number analyzed (Participants) | 8 | 11
  C2D21 | 27.0 [9 to 86] | 38.0 [8 to 141]
  C2D28: number analyzed (Participants) | 5 | 6
  C2D28 | 68.0 [48 to 333] | 173.0 [32 to 479]
  C2D35: number analyzed (Participants) | 2 | 3
  C2D35 | 515.0 [412 to 618] | 272.0 [26 to 329]
  C2D42: number analyzed (Participants) | 0 | 2
  C2D42 |  | 147.5 [45 to 250]

32. Secondary Outcome: Maximum Duration (Days) of Platelet Transfusion Independence
Description: Maximum time period (in days) during which the patient did not receive any platelet transfusion
Time Frame: At differnt time points from start of treatment and up to end of study year 2 assessment
Population: as for outcome 27
Measure: Median (Full Range); unit: Days
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 74
Days | 29.0 [2 to 57] | 29.5 [2 to 77]
Statistical Analysis 1: Comparison: Eltrombopag (ELQ) QD vs Placebo QD; Test type: Superiority; p = 0.6942, Wilcoxon rank-sum test

33. Secondary Outcome: Percentage of Patients Who Achieved Platelet Transfusion Independence ≥ 28 Days
Description: Percentage of patients who achieved platelet transfusion independence ≥ 28 days.
Time Frame: From start of treatment and up to end of study year 2 assessment
Population: as for outcome 27
Measure: Number; unit: Percentage of participants
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 74
Percentage of participants | 55 | 53
Statistical Analysis 1: Comparison: Eltrombopag (ELQ) QD vs Placebo QD; Test type: Superiority; p = 0.7397, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.1151, 95% CI 2-sided [0.5585 to 2.2290]

34. Secondary Outcome: Time to Neutrophil Engraftment
Description: Time to absolute neutrophil count (ANC) >= 0.5 Gi/L for 3 consecutive days in participants with ANC < 0.5 Gi/L after chemotherapy
Time Frame: At different time points from last dose of chemotherapy up to end of study year 2 assessment
Population: as for outcome 27
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 73
Months | NA [NA to NA] — N/A = Not enough participants achieved ANC>= 0.5 Gi/L | NA [NA to NA] — N/A = Not enough participants achieved ANC>= 0.5 Gi/L
Statistical Analysis 1: Comparison: Eltrombopag (ELQ) QD vs Placebo QD; Test type: Superiority; p = 0.0781, Log Rank; Hazard Ratio (HR) = 2.46, 95% CI 2-sided [0.95 to 6.38]

35. Secondary Outcome: Summary of Absolute Neutrophil Counts (ANC)
Description: Absolute neutrophil counts over time
Time Frame: as for outcome 31
Population: as for outcome 27
Measure: Median (Full Range); unit: Gi/L
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 74
Gi/L
  Baseline: number analyzed (Participants) | 71 | 72
  Baseline | 0.8 [0 to 37] | 0.5 [0 to 50]
  C1D1: number analyzed (Participants) | 55 | 63
  C1D1 | 0.8 [0 to 37] | 0.6 [0 to 50]
  C1D2: number analyzed (Participants) | 70 | 72
  C1D2 | 0.6 [0 to 41] | 0.5 [0 to 41]
  C1D3: number analyzed (Participants) | 66 | 70
  C1D3 | 0.6 [0 to 59] | 0.4 [0 to 26]
  C1D4: number analyzed (Participants) | 70 | 64
  C1D4 | 0.4 [0 to 35] | 0.2 [0 to 17]
  C1D5: number analyzed (Participants) | 70 | 63
  C1D5 | 0.3 [0 to 21] | 0.2 [0 to 2]
  C1D6: number analyzed (Participants) | 68 | 63
  C1D6 | 0.2 [0 to 35] | 0.1 [0 to 1]
  C1D7: number analyzed (Participants) | 69 | 62
  C1D7 | 0.1 [0 to 29] | 0.1 [0 to 1]
  C1D8: number analyzed (Participants) | 66 | 58
  C1D8 | 0.1 [0 to 21] | 0.0 [0 to 1]
  C1D9: number analyzed (Participants) | 66 | 59
  C1D9 | 0.0 [0 to 7] | 0.0 [0 to 1]
  C1D14: number analyzed (Participants) | 61 | 56
  C1D14 | 0.0 [0 to 1] | 0.0 [0 to 0]
  C1D21: number analyzed (Participants) | 52 | 51
  C1D21 | 0.6 [0 to 18] | 0.3 [0 to 7]
  C1D28: number analyzed (Participants) | 37 | 29
  C1D28 | 4.3 [0 to 47] | 2.7 [0 to 25]
  C1D35: number analyzed (Participants) | 14 | 14
  C1D35 | 2.2 [0 to 56] | 1.7 [0 to 12]
  C1D42: number analyzed (Participants) | 0 | 1
  C1D42 |  | 3.1 [3.1 to 3.1]
  C2D1: number analyzed (Participants) | 10 | 9
  C2D1 | 0.1 [0 to 7] | 0.0 [0 to 5]
  C2D2: number analyzed (Participants) | 10 | 9
  C2D2 | 0.1 [0 to 3] | 0.2 [0 to 4]
  C2D3: number analyzed (Participants) | 9 | 8
  C2D3 | 0.2 [0 to 5] | 0.5 [0 to 4]
  C2D4: number analyzed (Participants) | 9 | 9
  C2D4 | 0.3 [0 to 3] | 0.5 [0 to 2]
  C2D5: number analyzed (Participants) | 10 | 10
  C2D5 | 0.2 [0 to 2] | 0.1 [0 to 3]
  C2D6: number analyzed (Participants) | 10 | 10
  C2D6 | 0.1 [0 to 1] | 0.1 [0 to 3]
  C2D7: number analyzed (Participants) | 9 | 8
  C2D7 | 0.0 [0 to 1] | 0.1 [0 to 2]
  C2D14: number analyzed (Participants) | 7 | 8
  C2D14 | 0.0 [0 to 0] | 0.0 [0 to 0]

36. Secondary Outcome: Summary of Hemoglobin
Description: Hemoglobin level over time
Time Frame: as for outcome 31
Population: as for outcome 27
Measure: Median (Full Range); unit: g/L
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 74
g/L
  Baseline | 87.6 [63 to 123] | 87.0 [67 to 121]
  C1D1: number analyzed (Participants) | 60 | 66
  C1D1 | 88.0 [67 to 123] | 86.0 [67 to 121]
  C1D2 | 88.0 [58 to 124] | 83.0 [62 to 130]
  C1D3: number analyzed (Participants) | 74 | 72
  C1D3 | 86.0 [52 to 108] | 82.0 [59 to 130]
  C1D4: number analyzed (Participants) | 74 | 70
  C1D4 | 83.0 [60 to 105] | 81.5 [46 to 120]
  C1D5: number analyzed (Participants) | 74 | 71
  C1D5 | 84.0 [60 to 114] | 83.0 [50 to 126]
  C1D6: number analyzed (Participants) | 74 | 70
  C1D6 | 86.0 [67 to 118] | 82.0 [52 to 119]
  C1D7: number analyzed (Participants) | 74 | 71
  C1D7 | 85.0 [58 to 116] | 83.0 [57 to 110]
  C1D8: number analyzed (Participants) | 74 | 70
  C1D8 | 85.3 [65 to 118] | 84.0 [57 to 108]
  C1D9: number analyzed (Participants) | 74 | 70
  C1D9 | 84.5 [64 to 114] | 81.5 [62 to 109]
  C1D14: number analyzed (Participants) | 68 | 68
  C1D14 | 85.0 [60 to 123] | 84.0 [59 to 109]
  C1D21: number analyzed (Participants) | 52 | 55
  C1D21 | 88.0 [77 to 117] | 88.0 [72 to 116]
  C1D28: number analyzed (Participants) | 37 | 29
  C1D28 | 99.0 [78 to 138] | 98.0 [79 to 125]
  C1D35: number analyzed (Participants) | 14 | 14
  C1D35 | 99.0 [81 to 131] | 94.0 [74 to 130]
  C1D42: number analyzed (Participants) | 0 | 1
  C1D42 |  | 98.0 [98 to 98]
  C2D1: number analyzed (Participants) | 10 | 12
  C2D1 | 94.5 [76 to 124] | 82.5 [72 to 111]
  C2D2: number analyzed (Participants) | 10 | 12
  C2D2 | 88.5 [72 to 112] | 86.5 [69 to 104]
  C2D3: number analyzed (Participants) | 10 | 12
  C2D3 | 86.5 [65 to 110] | 80.0 [68 to 97]
  C2D4: number analyzed (Participants) | 10 | 12
  C2D4 | 89.0 [72 to 106] | 86.5 [74 to 109]
  C2D5: number analyzed (Participants) | 10 | 12
  C2D5 | 88.0 [67 to 101] | 84.0 [72 to 93]
  C2D6: number analyzed (Participants) | 10 | 12
  C2D6 | 84.0 [68 to 102] | 85.0 [70 to 96]
  C2D7: number analyzed (Participants) | 10 | 12
  C2D7 | 84.5 [66 to 99] | 83.0 [57 to 97]
  C2D14: number analyzed (Participants) | 11 | 8
  C2D14 | 77.5 [66 to 101] | 87.0 [79 to 96]
  C2D21: number analyzed (Participants) | 11 | 8
  C2D21 | 86.0 [43 to 99] | 91.0 [74 to 110]
  C2D28: number analyzed (Participants) | 7 | 5
  C2D28 | 89.0 [80 to 92] | 80.0 [72 to 114]
  C2D35: number analyzed (Participants) | 3 | 2
  C2D35 | 104.0 [101 to 107] | 87.0 [85 to 119]
  C2D42: number analyzed (Participants) | 0 | 2
  C2D42 |  | 90.5 [86 to 95]

37. Secondary Outcome: Incidence of Hemorrhagic Events
Description: Incidence of bleeding events using WHO bleeding grade (G0=No bleeding, G1=Petechiae, G2=Mild blood loss, G3=Gross blood loss, G4=Debilitating blood loss) by week and cycle
Time Frame: Baseline, weekly within induction and re-induction cycles, end of therapy
Population: as for outcome 27
Measure: Number; unit: Participants
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 74
Participants
  C1D7 - GRADE 0: number analyzed (Participants) | 73 | 69
  C1D7 - GRADE 0 | 58 | 47
  C1D7 - GRADE 1: number analyzed (Participants) | 73 | 69
  C1D7 - GRADE 1 | 9 | 16
  C1D7 - GRADE 2: number analyzed (Participants) | 73 | 69
  C1D7 - GRADE 2 | 5 | 6
  C1D7 - GRADE 3: number analyzed (Participants) | 73 | 69
  C1D7 - GRADE 3 | 1 | 0
  C1D14 - GRADE 0: number analyzed (Participants) | 68 | 65
  C1D14 - GRADE 0 | 42 | 43
  C1D14 - GRADE 1: number analyzed (Participants) | 68 | 65
  C1D14 - GRADE 1 | 16 | 13
  C1D14 - GRADE 2: number analyzed (Participants) | 68 | 65
  C1D14 - GRADE 2 | 5 | 6
  C1D14 - GRADE 3: number analyzed (Participants) | 68 | 65
  C1D14 - GRADE 3 | 1 | 0
  C1D21 - GRADE 0: number analyzed (Participants) | 52 | 52
  C1D21 - GRADE 0 | 36 | 43
  C1D21 - GRADE 1: number analyzed (Participants) | 52 | 52
  C1D21 - GRADE 1 | 13 | 7
  C1D21 - GRADE 2: number analyzed (Participants) | 52 | 52
  C1D21 - GRADE 2 | 3 | 1
  C1D21 - GRADE 3: number analyzed (Participants) | 52 | 52
  C1D21 - GRADE 3 | 0 | 1
  C1D28 - GRADE 0: number analyzed (Participants) | 37 | 28
  C1D28 - GRADE 0 | 31 | 25
  C1D28 - GRADE 1: number analyzed (Participants) | 37 | 28
  C1D28 - GRADE 1 | 4 | 3
  C1D28 - GRADE 2: number analyzed (Participants) | 37 | 28
  C1D28 - GRADE 2 | 2 | 0
  C1D28 - GRADE 3: number analyzed (Participants) | 37 | 28
  C1D28 - GRADE 3 | 0 | 0
  C1D35 - GRADE 0: number analyzed (Participants) | 14 | 13
  C1D35 - GRADE 0 | 12 | 11
  C1D35 - GRADE 1: number analyzed (Participants) | 14 | 13
  C1D35 - GRADE 1 | 2 | 2
  C1D35 - GRADE 2: number analyzed (Participants) | 14 | 13
  C1D35 - GRADE 2 | 0 | 0
  C1D35 - GRADE 3: number analyzed (Participants) | 14 | 13
  C1D35 - GRADE 3 | 0 | 0
  C1D42 - GRADE 0: number analyzed (Participants) | 0 | 1
  C1D42 - GRADE 0 |  | 0
  C1D42 - GRADE 1: number analyzed (Participants) | 0 | 1
  C1D42 - GRADE 1 |  | 1
  C1D42 - GRADE 2: number analyzed (Participants) | 0 | 1
  C1D42 - GRADE 2 |  | 0
  C1D42 - GRADE 3: number analyzed (Participants) | 0 | 1
  C1D42 - GRADE 3 |  | 0
  C2D1 - GRADE 0: number analyzed (Participants) | 10 | 12
  C2D1 - GRADE 0 | 8 | 8
  C2D1 - GRADE 1: number analyzed (Participants) | 10 | 12
  C2D1 - GRADE 1 | 1 | 4
  C2D1 - GRADE 2: number analyzed (Participants) | 10 | 12
  C2D1 - GRADE 2 | 1 | 0
  C2D1 - GRADE 3: number analyzed (Participants) | 10 | 12
  C2D1 - GRADE 3 | 0 | 0
  C2D7 - GRADE 0: number analyzed (Participants) | 10 | 11
  C2D7 - GRADE 0 | 9 | 8
  C2D7 - GRADE 1: number analyzed (Participants) | 10 | 11
  C2D7 - GRADE 1 | 0 | 3
  C2D7 - GRADE 2: number analyzed (Participants) | 10 | 11
  C2D7 - GRADE 2 | 1 | 0
  C2D7 - GRADE 3: number analyzed (Participants) | 10 | 11
  C2D7 - GRADE 3 | 0 | 0
  C2D14 - GRADE 0: number analyzed (Participants) | 8 | 10
  C2D14 - GRADE 0 | 8 | 7
  C2D14 - GRADE 1: number analyzed (Participants) | 8 | 10
  C2D14 - GRADE 1 | 0 | 3
  C2D14 - GRADE 2: number analyzed (Participants) | 8 | 10
  C2D14 - GRADE 2 | 0 | 0
  C2D14 - GRADE 3: number analyzed (Participants) | 8 | 10
  C2D14 - GRADE 3 | 0 | 0
  C2D21 - GRADE 0: number analyzed (Participants) | 8 | 9
  C2D21 - GRADE 0 | 7 | 7
  C2D21 - GRADE 1: number analyzed (Participants) | 8 | 9
  C2D21 - GRADE 1 | 1 | 2
  C2D21 - GRADE 2: number analyzed (Participants) | 8 | 9
  C2D21 - GRADE 2 | 0 | 0
  C2D21 - GRADE 3: number analyzed (Participants) | 8 | 9
  C2D21 - GRADE 3 | 0 | 0
  C2D28 - GRADE 0: number analyzed (Participants) | 5 | 8
  C2D28 - GRADE 0 | 5 | 7
  C2D28 - GRADE 1: number analyzed (Participants) | 5 | 8
  C2D28 - GRADE 1 | 0 | 1
  C2D28 - GRADE 2: number analyzed (Participants) | 5 | 8
  C2D28 - GRADE 2 | 0 | 0
  C2D28 - GRADE 3: number analyzed (Participants) | 5 | 8
  C2D28 - GRADE 3 | 0 | 0
  C2D35 - GRADE 0: number analyzed (Participants) | 3 | 3
  C2D35 - GRADE 0 | 3 | 2
  C2D35 - GRADE 1: number analyzed (Participants) | 3 | 3
  C2D35 - GRADE 1 | 0 | 1
  C2D35 - GRADE 2: number analyzed (Participants) | 3 | 3
  C2D35 - GRADE 2 | 0 | 0
  C2D35 - GRADE 3: number analyzed (Participants) | 3 | 3
  C2D35 - GRADE 3 | 0 | 0
  C2D42 - GRADE 0: number analyzed (Participants) | 0 | 1
  C2D42 - GRADE 0 |  | 0
  C2D42 - GRADE 1: number analyzed (Participants) | 0 | 1
  C2D42 - GRADE 1 |  | 1
  C2D42 - GRADE 2: number analyzed (Participants) | 0 | 1
  C2D42 - GRADE 2 |  | 0
  C2D42 - GRADE 3: number analyzed (Participants) | 0 | 1
  C2D42 - GRADE 3 |  | 0
  Remission visit GRADE 0: number analyzed (Participants) | 62 | 62
  Remission visit GRADE 0 | 56 | 58
  Remission visit GRADE 1: number analyzed (Participants) | 62 | 62
  Remission visit GRADE 1 | 2 | 4
  Remission visit GRADE 2: number analyzed (Participants) | 62 | 62
  Remission visit GRADE 2 | 3 | 0
  Remission visit GRADE 3: number analyzed (Participants) | 62 | 62
  Remission visit GRADE 3 | 1 | 0

38. Secondary Outcome: Percentage of Participants With Disease Response Rate and Type of Response
Description: Disease response as assessed by the investigator using the AML International Working Group Response Assessment at the end of therapy/remission assessment visit; Complete remission (CR): defined as transfusion independence, blood count recovery (Abs. neutrophil count > 1.0 Gi/L and Platelet count > 100.0 Gi/L), no leukemic blast in peripheral blood, Bone Marrow (BM) blasts < 5%, maturation of all cell lines, Auer rods not detectable, and no extramedullary disease.
  Partial remission (PR): defined as CR except that for BM blasts where a decrease of at least 50% of BM blasts to 5-25% in BM aspirate is sufficient or BM blasts < 5% with Auer rods present.
  Overall response (OR) = CR + PR.
Time Frame: Day 42 of the latest chemotherapy cycle (Up to 8 weeks)
Population: as for outcome 27
Measure: Number; unit: Percentage of participants
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 74
Percentage of participants
  Overall response | 70 | 73
  Complete Remission (CR) | 65 | 70
  Partial Remission (PR) | 5 | 3
Statistical Analysis 1: Comparison: Eltrombopag (ELQ) QD vs Placebo QD; Test type: Superiority; p = 0.7122, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.8749, 95% CI 2-sided [0.4023 to 1.8943]

39. Secondary Outcome: Overall Survival (OS)
Description: Overall survival defined as the time form randomization until the date of death due to any cause.
Time Frame: From randomization to end of 2-year follow-up
Population: as for outcome 27
Measure: Number; unit: Count of participants
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 74
Count of participants | 39 | 30
Statistical Analysis 1: Comparison: Eltrombopag (ELQ) QD vs Placebo QD; Test type: Superiority; p = 0.0688, Log Rank; Hazard Ratio (HR) = 1.54, 95% CI 2-sided [0.96 to 2.47]

40. Secondary Outcome: Number of Participants Who Required Medical Resource Utilization
Description: Medical Resource Utilization pertained to unscheduled hospitalizations, unscheduled office visits, unscheduled laboratory tests, and unscheduled procedures.
Time Frame: At screening and from start of treatment to end of therapy/remission assessment visit (Day 42 of the latest chemotherapy cycle)
Population: as for outcome 27
Measure: Number; unit: Count of participants
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
Number analyzed (Participants) | 74 | 74
Count of participants
  In-patient hospitalizations/ admissions? | 3 | 4
  Diagnostic imaging procedures performed? | 3 | 4
  Health care resources use or emergency visits? | 8 | 6
  Out-patient lab tests performed? | 6 | 6

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected from Day 1 of cycle 1 until last dose of investigational product + 30 days i.e. a maximum of 114 days (42 days for the induction cycle + 42 days for the re-induction cycle + 30 days for the follow-up)
Arm/Group | Eltrombopag (ELQ) QD | Placebo QD
All-Cause Mortality (participants affected / at risk) | 11/74 | 4/71
Serious Adverse Events (participants affected / at risk) | 24/74 | 14/71
Other Adverse Events (participants affected / at risk) | 71/74 | 66/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (ELQ) QD (N=74) | Placebo QD (N=71)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1
Generalised oedema (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Sudden death (General disorders) | 0 | 1
Acinetobacter bacteraemia (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 1
Klebsiella sepsis (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 2
Septic shock (Infections and infestations) | 2 | 2
Systemic candida (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Pseudohyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (ELQ) QD (N=74) | Placebo QD (N=71)
Anaemia (Blood and lymphatic system disorders) | 7 | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 38 | 42
Neutropenia (Blood and lymphatic system disorders) | 5 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 4
Thrombocytosis (Blood and lymphatic system disorders) | 5 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 4
Abdominal discomfort (Gastrointestinal disorders) | 2 | 4
Abdominal distension (Gastrointestinal disorders) | 2 | 6
Abdominal pain (Gastrointestinal disorders) | 18 | 17
Abdominal pain lower (Gastrointestinal disorders) | 0 | 4
Abdominal pain upper (Gastrointestinal disorders) | 3 | 12
Constipation (Gastrointestinal disorders) | 28 | 21
Diarrhoea (Gastrointestinal disorders) | 42 | 43
Dry mouth (Gastrointestinal disorders) | 7 | 2
Dyspepsia (Gastrointestinal disorders) | 10 | 9
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 4
Gingival bleeding (Gastrointestinal disorders) | 6 | 4
Gingival pain (Gastrointestinal disorders) | 4 | 3
Gingival swelling (Gastrointestinal disorders) | 3 | 5
Haemorrhoids (Gastrointestinal disorders) | 10 | 9
Lip dry (Gastrointestinal disorders) | 4 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 5 | 0
Mouth ulceration (Gastrointestinal disorders) | 2 | 4
Nausea (Gastrointestinal disorders) | 37 | 46
Proctalgia (Gastrointestinal disorders) | 4 | 10
Stomatitis (Gastrointestinal disorders) | 19 | 18
Vomiting (Gastrointestinal disorders) | 27 | 27
Asthenia (General disorders) | 13 | 13
Catheter site haemorrhage (General disorders) | 4 | 1
Chest pain (General disorders) | 0 | 4
Chills (General disorders) | 21 | 14
Fatigue (General disorders) | 10 | 11
Mucosal inflammation (General disorders) | 9 | 9
Oedema (General disorders) | 6 | 6
Oedema peripheral (General disorders) | 12 | 13
Pain (General disorders) | 3 | 6
Pyrexia (General disorders) | 25 | 17
Bacteraemia (Infections and infestations) | 4 | 1
Cellulitis (Infections and infestations) | 0 | 6
Device related infection (Infections and infestations) | 6 | 9
Oral candidiasis (Infections and infestations) | 1 | 6
Pneumonia (Infections and infestations) | 8 | 3
Sepsis (Infections and infestations) | 5 | 3
Procedural pain (Injury, poisoning and procedural complications) | 5 | 5
Transfusion reaction (Injury, poisoning and procedural complications) | 10 | 8
Alanine aminotransferase increased (Investigations) | 8 | 14
Aspartate aminotransferase increased (Investigations) | 5 | 8
Blood bilirubin increased (Investigations) | 6 | 8
Neutrophil count decreased (Investigations) | 4 | 1
Platelet count decreased (Investigations) | 7 | 4
Serum ferritin increased (Investigations) | 6 | 2
Weight increased (Investigations) | 1 | 5
White blood cell count decreased (Investigations) | 9 | 5
Decreased appetite (Metabolism and nutrition disorders) | 22 | 27
Fluid imbalance (Metabolism and nutrition disorders) | 12 | 10
Fluid overload (Metabolism and nutrition disorders) | 6 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 7 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 20 | 27
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 | 13
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 10 | 14
Iron overload (Metabolism and nutrition disorders) | 6 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 15
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 8
Dizziness (Nervous system disorders) | 11 | 8
Headache (Nervous system disorders) | 19 | 20
Anxiety (Psychiatric disorders) | 10 | 7
Insomnia (Psychiatric disorders) | 16 | 23
Haematuria (Renal and urinary disorders) | 1 | 4
Urinary hesitation (Renal and urinary disorders) | 5 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 18 | 14
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 | 13
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 4
Erythema (Skin and subcutaneous tissue disorders) | 5 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 12 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 8
Rash (Skin and subcutaneous tissue disorders) | 22 | 13
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 | 6
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 4
Hypertension (Vascular disorders) | 6 | 8
Hypotension (Vascular disorders) | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety